CLINICAL TRIAL: NCT06609811
Title: The Interaction Between Mucosal Microbiota Colonization in the Nasal Cavity and Gut and the Immune Response to an Intranasal Influenza Live Attenuated Vaccine in Children and Adolescents Aged 6 to 17 Years: A Single-Center, Randomized, Open-Label Trial
Brief Title: The Interaction Between Mucosal Microbiota Colonization and the Immune Response to an Intranasal Influenza Live Attenuated Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSJKYMS001
Record Dates: First submitted 2024-09-13; First posted 2024-09-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Influenza
Keywords: Intranasal Influenza Live Attenuated Vaccine; Nasal Microbiota; Gut Microbiota; Colonization; Mucosal Immunity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The immediate vaccination group. (Experimental): Participants are assigned to receive one dose of 0.2 mL of intranasal live attenuated influenza vaccine immediately (Day 0)
  Interventions: Biological: Intranasal Influenza Live Attenuated Vaccine
- The delayed vaccination group (Experimental): Participants are assigned to receive one dose of 0.2 mL of intranasal live attenuated influenza vaccine after a delay (Day 28).
  Interventions: Biological: Intranasal Influenza Live Attenuated Vaccine

INTERVENTIONS:
Biological: Intranasal Influenza Live Attenuated Vaccine — This vaccine is produced by Changchun BCHT Biotechnology Co.
  Arms: The delayed vaccination group
Biological: Intranasal Influenza Live Attenuated Vaccine — This vaccine is produced by Changchun BCHT Biotechnology Co.
  Arms: The immediate vaccination group.

SUMMARY:
This is a single-center, randomized, open-label trial designed to explore the interaction between mucosal microbiota colonization in the nasal cavity and gut and the immune response to an intranasal live attenuated influenza vaccine (LAIV). The study plans to enroll 200 children and adolescents aged 6-17 years, with approximately 50% in the 6-11 years age group and 50% in the 12-17 years age group. Participants and their guardians must be able and willing to comply with the clinical trial protocol and provide informed consent. Eligible participants will be randomly assigned in a 1:1 ratio, stratified by age groups, to either the immediate vaccination group or the delayed vaccination group. Nasal swabs will be collected for all participants of both the immediate vaccination group or the delayed vaccination group after randomization for the detection of nasal and gut microbiota. Then, the immediate vaccination group will receive one dose of 0.2 mL of LAIV 28 days after randomization, while the delayed vaccination group will receive one dose of 0.2 mL of LAIV 56 days after randomization. Blood and mucosal samples (nasal stool) will be collected on the day before vaccination and on 28 days after vaccination for humoral and mucosal immunogenicity analysis. Moreover, the occurrence of adverse events within 28 days after vaccination will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 6-17 years.
2. Volunteers and their guardians are able and willing to comply with the requirements of the clinical trial protocol and sign the informed consent form.

Exclusion Criteria:

1. Allergy to any component of the vaccine product, including eggs, excipients, or gentamicin sulfate.
2. Individuals with acute illnesses, severe chronic illnesses, acute exacerbations of chronic illnesses, or fever.
3. Pregnant or lactating women.
4. Individuals with Leigh syndrome who are receiving treatment with aspirin or aspirin-containing medications.
5. Individuals with immunodeficiency, immunosuppression, or those undergoing immunosuppressive therapy.
6. Individuals with uncontrolled epilepsy, other progressive neurological disorders, or a history of Guillain-Barré syndrome.
7. Individuals with rhinitis or asthma.
8. Individuals with a personal or family history of seizures, chronic diseases, epilepsy, or allergic tendencies.
9. Individuals who have received immunoglobulin injections within the last 3 months prior to vaccination.
10. Individuals who have used other live attenuated vaccines within 1 month prior to vaccination.
11. Individuals planning to use antiviral drugs for influenza within 48 hours before or 2 weeks after vaccination.
12. Individuals planning to use any other intranasal medication within 2 days after vaccination.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
The level of sIgA antibodies (ng/mL) against the vaccine strain in nasal secretions at 28 days post-vaccination | Day 28 post-vaccination
  Measured by Meso Scale Discovery
Changes in the density of nasal mucosal bacterial colonization (CFU/mL) compared to baseline | Day 28 post-vaccination
  Measured by 16s RNA or metagenomic analysis
Changes in the abundance (α Diversity and β Diversity) of nasal mucosal bacterial colonization compared to baseline | Day 28 post-vaccination
  Measured by 16s RNA or metagenomic analysis

SECONDARY OUTCOMES:
The level of neutralizing antibodies (NT50 and IC50, ng/mL) against the vaccine strain in serum at 28 days post-vaccination | Day 28 post-vaccination
  Measured by Neutralization Assay
Changes in the density of gut bacterial colonization (CFU/mL) compared to baseline | Day 28 post-vaccination
  Measured by 16s RNA or metagenomic analysis
Changes in the abundance (α Diversity and β Diversity) of gut bacterial colonization compared to baseline | Day 28 post-vaccination
  Measured by 16s RNA or metagenomic analysis
The incidence of adverse events (AEs) within 28 days post-vaccination | within 28 days post-vaccination
Number of IFN-γ secreting cells in nasal mucosal epithelial cells in response to influenza virus-based synthetic peptide pools at Day 28 post-vaccination (Exploratory) | Day 28 post-vaccination
  The number of IFN-γ secreting cells will be quantified using an ELISpot assay.
Frequency of activated T-cell subsets in nasal mucosal epithelial cells at Day 28 post-vaccination (Exploratory) | Day 28 post-vaccination
  The phenotype and activation status of local mucosal T-cell subsets were measured by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention; Jiangsu Provincial Center for Diseases Control and Prevention, Study Director — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Haizhou District Center for Disease Control and Prevention, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No